CLINICAL TRIAL: NCT05457933
Title: Efficacy and Safety of Dapagliflozin for the Hospital Management of Patients With Type 2 Diabetes: a Prospective, Open-label, Non-inferiority Randomized Trial
Brief Title: Efficacy and Safety of Dapagliflozin for the Hospital Management of Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medanta, The Medicity, India (Other)
Responsible Party: Principal Investigator, Dr Mohammad Shafi Kuchay, Consultant, Medanta, The Medicity, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMDAPHS01
Record Dates: First submitted 2022-07-05; First posted 2022-07-14 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Type2diabetes; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — dapagliflozin; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin group (Experimental): Dapagliflozin 10 mg, every day before breakfast. Glargine insulin 300 Units/mL, average dose: 10-20 U/day; Insulin lispro 100 Units/mL, average dose: 10-30 U/day
  Interventions: Drug: Dapagliflozin
- Basal-bolus group (Active Comparator): Glargine insulin; 300 Units/mL, average dose: 10-20 U/day; Insulin lispro 100 Units/mL, average dose: 10-30 U/day
  Interventions: Drug: Glargine

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg, every day before breakfast. Glargine insulin 300 Units/mL, average dose: 10-20 U/day; Insulin lispro 100 Units/mL, average dose: 10-30 U/day
  Arms: Dapagliflozin group
Drug: Glargine — Glargine insulin; 300 Units/mL, average dose: 10-20 U/day, Insulin lispro 100 Units/mL, average dose: 10-30 U/day
  Other Names: Lispro
  Arms: Basal-bolus group

SUMMARY:
The purpose of the trial is to examine whether treatment with dapagliflozin plus insulin as compared with insulin alone (basal-bolus insulin) will result in similar blood glucose control and similar rate of complications in patients with diabetes, who are admitted to a hospital in a noncritical setting

DETAILED DESCRIPTION:
Background

Good glycemic control is crucial for improving clinical outcomes in hospitalized patients with diabetes. Multiple insulin injections (one dose of long-acting insulin and three doses of rapid-acting pre-meal bolus insulins) are the standard of care for the hospital management of patients with diabetes. Sodium-glucose cotransporter 2 (SGLT-2) inhibitors is a class of glucose-lowering agents that are increasingly being used in patients with type 2 diabetes, due to multiple pleiotropic effects. These drugs reduce cardiovascular mortality, especially by reducing risk of heart failure, and also improve renal outcomes. The role of SGLT-2 inhibitors in the treatment of patients admitted to hospital in a non-critical care setting has not been assessed. Accordingly, the proposed study will provide a clinically useful information on the efficacy (blood glucose control) and safety (hypoglycemia) of dapagliflozin (an SGLT-2 inhibitor) for the management of hospitalized patients with type 2 diabetes.

Summary

The purpose of the trial is to examine whether treatment with dapagliflozin plus insulin as compared with insulin alone (basal-bolus insulin) will result in similar blood glucose control and similar rate of complications in patients with diabetes, who are admitted to a hospital in a noncritical setting.

Arms and interventions

Arms Study participants with type 2 diabetes undergoing elective coronary artery bypass graft (CABG) surgery will receive basal-bolus regimen (one dose of long-acting basal insulin and three doses of rapid-acting pre-meal bolus insulins) on the third day of surgery (transition from intravenous insulin infusion). One arm (dapagliflozin group) will receive dapagliflozin 10 mg daily in addition to basal-bolus regimen while another group (basal-bolus group) will receive basal-bolus insulin without dapagliflozin. Both arms will receive glargine U300 as basal insulin and lispro U100 as rapid-acting bolus insulin.

Dapagliflozin group:

Dapagliflozin 10 mg, every day before breakfast. Glargine insulin 300 Units/mL, average dose: 10-20 U/day; Insulin lispro 100 Units/mL, average dose: 10-30 U/day

Basal-bolus group:

Glargine insulin; 300 Units/mL, average dose: 10-20 U/day; Insulin lispro 100 Units/mL, average dose: 10-30 U/day

Primary outcome measure Noninferiority in mean differences between groups in their daily blood glucose concentrations. [Time Frame: The first 7 days of therapy in hospital and 5 days post-discharge]

Blood glucose will be measured pre-breakfast, pre-lunch, pre-dinner and night-time (0300 hours). Mean daily blood glucose concentration will be calculated to determine differences in inpatient glycemic control in patients with type 2 diabetes treated with dapagliflozin 10 mg plus basal-bolus insulin or basal-bolus regimen, using glargine U300 as basal insulin and insulin lispro U100 before meals.

Sample size calculation

Noninferiority for the primary end point of glycemic control will be defined as a mean blood glucose difference of <18 mg/dL between dapagliflozin group and basal-bolus group. A blood glucose difference of such a magnitude has been reported in other superiority trials as nonclinically significant and is smaller than significant treatment effects. Assuming the true blood glucose difference between the treatment groups is zero, and using one-sided, two-sample t tests, Principal Investigato required 90 subjects for each treatment group to achieve 90% power. Principal Investigator do not expect any attrition rate. Principal Investigato aimed to enrol 200 subjects in total to achieve >90% power.

Procedures

Patients will be treated with a basal-bolus insulin regimen approach as previously reported. In brief, all study participants will receive insulin infusion till soft diet is initiated. Dose of insulin (units/hour) for last 4 hours will be calculated and that dose will be multiplied by 24 to get the 24 hour insulin utilization, and 80% of that 24-h dose was be as total daily dose (TDD). Half of the TDD will be administered as once-daily basal insulin (glargine U300) at 11:00 am, and half as prandial insulin (lispro U100) divided in three equal doses before meals. Insulin infusion will be continued till lunch time, and will be discontinued once pre-lunch rapid-acting bolus dose is administered. No interim analysis will be performed. Dapagliflozin group will receive first dose of dapagliflozin 10 mg, before lunch on the same day, followed by before breakfast next day onwards.

Glargine U100 will be given once daily, at the same time of the day (11:00 am). Insulin doses will be adjusted daily to maintain a fasting blood glucose <140 mg/dL, and pre-meals <180 mg/dL, while avoiding hypoglycemia <70 mg/dL. The TDD will be increased by 10% if blood glucose was between 140 and 180 mg/dL, by 20% if BG was between 180 and 240 mg/dL, and by 30% if BG was >240 mg/dL.

Glucose Monitoring

Glucose levels will be assessed by capillary point-of-care (POC) testing before meals, and at night-time (0300 hours). A subgroup of participants (n = 100) will wear a professional (blinded) Abbott FreeStyle Libre continuous glucose monitor (CGM).

Statistical Analysis

Noninferiority for the primary end point of glycemic control was defined as a mean BG difference of <18 mg/dL between dapagliflozin group and basal-bolus group. . A BG difference of such a magnitude has been reported in other superiority trials as nonclinically significant and is smaller than significant treatment effects. Assuming the true BG difference between the treatment groups is zero, and using one-sided, two-sample t tests, Principal Investigato required 90 participants for each treatment group to achieve 90% power. Accounting for a 5% attrition rate, Principal Investigatoaimed to enrol 200 participants in total to achieve >90% power. To compare baseline and clinical characteristics and outcomes, such as mean daily BG, occurrence of hypoglycemia, and occurrence of complications between treatment groups,Principal Investigato used nonparametric Wilcoxon tests for continuous variables and χ2 tests (or the Fisher exact test) for discrete variables. To determine differences in the primary end point, Principal Investigatoperformed a cross-sectional analysis using nonparametric Kruskal-Wallis tests (or Wilcoxon tests) or one-way ANOVA, followed by repeated-measures ANOVA to estimate and test the difference between the two treatment groups while simultaneously examining mean daily BG across multiple days during treatment. Secondary end point analysis was not adjusted for multiple comparisons. A P value of <0.05 was considered significant. The data are presented as mean ± SD for continuous variables and count (percentage) for discrete variables. Principal Investigatoperformed the statistical analyses with SAS 9.4 software.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females 30 years or above admitted to the hospital for elective CABG surgery
2. A known history of type 2 diabetes treated with any combination of oral antidiabetic agents, short-acting GLP1-RA (exenatide, liraglutide) or insulin therapy.
3. Study participants must have a randomization total daily dose (TDD) insulin requirement of at least 12 units per day.
4. Signed, informed consent prior to any study procedures

Exclusion Criteria:

1. Subjects with increased BG concentration, but without a known history of diabetes (stress hyperglycemia).
2. Subjects treated with diet alone (no antidiabetic agents) and admission HbA1c <7%.
3. Subjects with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria.
4. Patients treated with long-acting weekly GLP1-RA (weekly exenatide, or dulaglutide).
5. Any known hypersensitivity to dapagliflozin.
6. History of recurrent urinary tract infections (>2 episodes) requiring antibiotic therapy in the last 1 year.
7. History of intolerance to dapagliflozin or any other sodium-glucose cotransporter 2 inhibitors.
8. Patients with history of clinically relevant hepatic disease (diagnosed liver cirrhosis and portal hypertension).
9. Patients with ongoing corticosteroid therapy (equal to a prednisone dose ≥5 mg/day).
10. Patients with impaired renal function (eGFR <45 ml/min/1.73m2).
11. Patients with congestive heart failure (NYHA- IV).
12. Patients with medical and surgical pancreatic disease.
13. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
14. Body mass index (BMI) <18.5 kg/m2.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-01-14 (Actual); Study Completion 2023-01-14 (Actual)

PRIMARY OUTCOMES:
Noninferiority in mean differences between groups in their daily blood glucose concentrations | The first 7 days of therapy in hospital and 5 days post-discharge
  Blood glucose will be measured pre-breakfast, pre-lunch, pre-dinner and night-time (0300 hours). Mean daily blood glucose concentration will be calculated to determine differences in inpatient glycemic control in patients with type 2 diabetes treated with dapagliflozin 10 mg plus basal-bolus insulin or basal-bolus regimen, using glargine U300 as basal insulin and insulin lispro U100 before meals.

SECONDARY OUTCOMES:
Number of basic glucose readings between 70 mg/dl and 180 mg/dl before meals and night-time in hospitalized patients. | The first 7 days of therapy in hospital and 5 days post-discharge.
  Blood glucose will be measured before each meal and at night-time (0300 hours), and proportion of basic glucose readings between 70 mg/dl and 180 mg/dl will be recorded.
Number of hypoglycemic episodes (BG < 70 mg/dl and 54 mg/dl) in hospitalized patients. | The first 7 days of therapy in hospital and 5 days post-discharge.
  Blood glucose will be measured before each meal and at night-time (0300 hours), and number of hypoglycemic episodes (< 70 mg/dl and 54 mg/dl) will be recorded.
Number of severe hypoglycemia (< 54 mg/dl) episodes in hospitalized patients. | The first 7 days of therapy in hospital and 5 days post-discharge
  Blood glucose will be measured before each meal and at night-time (0300 hours, and number of hypoglycemia (< 54 mg/dl) episodes will be recorded.
Number of episodes of severe hyperglycemia (BG > 240 mg/dl) in hospitalized patients. | The first 7 days of therapy in hospital and 5 days post-discharge.
  Blood glucose will be measured before each meal and at night-time (0300 hours, and number of severe hyperglycemia (> 240 mg/dl) episodes will be recorded.
Daily dose of basal insulin, daily dose of prandial insulin, and total daily dose in hospitalized patients. | The first 7 days of therapy in hospital and 5 days post-discharge.
  The study team will document day and time of insulin administration of study drug given once daily and prandial- rapid-acting insulin (lispro U100) given before meals. The study team will also record dose and number of units given as supplement (correction) to correct hyperglycemia.
Continuous Glucose Monitoring | The first 7 days of therapy in hospital and 5 days post-discharge.
  Average blood glucose (mg/dL), percentage time in target (TIR), percentage time below target (TBR), and percentage time above target (TAR) in a subgroup of study participants using professional, blinded continuous glucose monitoring system (CGMS).
Hospital complications | The first 7 days of therapy in hospital and 5 days post-discharge.
  Hospital complications will be documented in all patients: complications like mortality, sternal wound infections, acute kidney injury, consolidation/pneumonia/pleural effusion, stroke and cardiac arrthymias.
Serum Ketone levels | Day 0, 3 and 5 of randomization
  Differences in number of patients who develop ketonemia. [Serum ketone body levels will be performed in all patients at day of randomization (day 0), day 3 and Day 5 of randomization.
Diabetic acidosis | The first 7 days of therapy in hospital and 5 days post-discharge.
  Differences in number of patients who develop acidosis. [Venous blood gas (VBG) assessment in all patients with ketonemia].
Glycated hemoglobin | 3 Months
  Glycated hemoglobin will be re-assessed at 3-month
Fasting blood glucose | 3 Months
  fasting blood glucose will be re-assessed at 3-month
Complete blood count | 3 Months
  Complete blood count will be re-complete blood count assessed at 3-month
Liver function test | 3 Months
  liver function test will be re-assessed at 3-month
Kidney function test | 3 Months
  kidney function test will be re-assessed at 3-month
A Composite of re-admission for heart failure or for any other reason | 3 Months
  Clinical complications namely re-admission for heart failure, or re-admission for any other reason will be re-assessed in all patients at 3-month.
Diuretics Use | 3 Months
  Dose of diuretics will be documented in all patients at 3-month.

CONTACTS AND LOCATIONS:
Locations (1):
- Division Of Endocrinology and Diabetes, Medanta The Medicity, Gurgaon, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pasquel FJ, Lansang MC, Dhatariya K, Umpierrez GE. Management of diabetes and hyperglycaemia in the hospital. Lancet Diabetes Endocrinol. 2021 Mar;9(3):174-188. doi: 10.1016/S2213-8587(20)30381-8. Epub 2021 Jan 27. PMID 33515493
- [Result] Damman K, Beusekamp JC, Boorsma EM, Swart HP, Smilde TDJ, Elvan A, van Eck JWM, Heerspink HJL, Voors AA. Randomized, double-blind, placebo-controlled, multicentre pilot study on the effects of empagliflozin on clinical outcomes in patients with acute decompensated heart failure (EMPA-RESPONSE-AHF). Eur J Heart Fail. 2020 Apr;22(4):713-722. doi: 10.1002/ejhf.1713. Epub 2020 Jan 7. PMID 31912605
- [Derived] Kuchay MS, Khatana P, Mishra M, Surendran P, Kaur P, Wasir JS, Gill HK, Singh A, Jain R, Kohli C, Bakshi G, Radhika V, Saheer S, Singh MK, Mishra SK. Dapagliflozin for inpatient hyperglycemia in cardiac surgery patients with type 2 diabetes: randomised controlled trial (Dapa-Hospital trial). Acta Diabetol. 2023 Nov;60(11):1481-1490. doi: 10.1007/s00592-023-02138-4. Epub 2023 Jun 29. PMID 37380728